CLINICAL TRIAL: NCT00062595
Title: Vitamin K and Bone Turnover in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Eisai Co., Ltd. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DK58363 (completed 2005)
Record Dates: First submitted 2003-06-09; First posted 2003-06-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Osteoporosis
Keywords: Menopause; Vitamin K; Bone turnover; Bone Density
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin K 1

INTERVENTIONS:
Drug: phylloquinone (K1)
Drug: menatetranone (MK4)

SUMMARY:
This one year study of the K vitamers phylloquinone (K1) and menatetranone (MK4) will study supplementation effects on bone turnover and bone density. Women at least 5 years postmenopause with normal bone density who do not use estrogen therapy or the following medications may be eligible:

alendronate (Fosamax), risedronate (Actonel), pamidronate (Aredia), etidronate (Didronel), zoledronate (Zometa), teriparatide (Forteo), raloxifene (Evista), tamoxifene, warfarin (Coumadin), anti-seizure medications, prednisone, or oral steroids. Eligible subjects will take calcium and vitamin D (Citracal) twice a day for the first two months and through-out the study. After the first two months, subjects are randomized to the K1, MK4 or placebo groups. Return visits occur at 1, 3, 6 and 12 months. Fasting blood and urine is collected at each visit and bone density is performed at 3 study visits.

ELIGIBILITY:
* Female, 5 years postmenopause.
* Ambulatory.
* Community dwelling.
* Able to ingest calcium and vitamin D supplements.
* Willing to restrict vitamin K intake.
* Stable thyroid dose if appropriate.
* No history of hyperthyroidism, hyperparathyroidism or other metabolic bone diseases.
* Absence of hardware in hip and spine.
* History of malignancy within the last five years.
* Not currently using coumadin or warfarin.
* Vitamin D supplements must be less than 800 IU daily.
* Have not used estrogen or other bone-altering medications (see list in study description) within the last year.
* No history of liver disease or malabsorption.
* No known allergy to vitamin K.
* Have not participated in an investigational drug trial within the last month.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 375
Dates: Start 2000-09; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin Osteoporosis Clinical Research Prog., Madison, Wisconsin, United States

REFERENCES:
- [Derived] Kumar R, Binkley N, Vella A. Effect of phylloquinone supplementation on glucose homeostasis in humans. Am J Clin Nutr. 2010 Dec;92(6):1528-32. doi: 10.3945/ajcn.2010.30108. Epub 2010 Sep 29. PMID 20881072